CLINICAL TRIAL: NCT06622837
Title: Within-subject Evaluation of Swallowing Threshold and Efficiency for Maxillary Implant Assisted Overdenture with and Without Palatal Coverage.
Brief Title: Swallowing Threshold and Efficiency for Maxillary Implant Assisted Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A0408024RP
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Prosthesis Durability
Keywords: Palatless,; Maxillary; Implant; Overdenture; swallowing
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I conventional maxillary implant overdenture (Active Comparator): Conventional MaxIOD: After relieving the conventional maxillary denture, direct pick-up technique was used to incorporate the attachments housing into the fitting surface of the conventional maxillary denture.
  Interventions: Procedure: implant overdenture
- group II palatless maxillary implant overdenture (Active Comparator): Palateless MaxIOD: The conventional maxillary denture was duplicated and the palatal part was cut out, finished, and polished. The fitting surface was relived and direct pick-up technique was used to incorporate the attachments housing into the fitting surface of the palateless maxillary denture.
  Interventions: Procedure: implant overdenture

INTERVENTIONS:
Procedure: implant overdenture — With the assistance of these stereolithographic surgical guides and submerged surgical technique, 4 dental implants (IS III Active Implant, Neo BioTech) were placed in the canines and premolars regions of the maxillary arch, and 2 dental implants were placed in the canines region of the mandibular arch.

SUMMARY:
This study aimed to compare the swallowing threshold and efficiency of conventional maxillary implant overdenture and palatless designs.

DETAILED DESCRIPTION:
New complete dentures were constructed for each participants using the conventional technique. The dentures were then inserted and adjusted according to a lingualized balanced occlusal scheme. The dentures were duplicated using clear acrylic resin material. Radiopaque gutta percha markers were placed on the labial, buccal, and lingual flanges of the clear resin duplicate at different axial planes to create a radiographic stent.

For each participant, dual scan was performed using cone beam computerized tomography ( i-CAT, Pennsylvania, USA). One scan was taken while the patient wore the radiographic stent, and the other scan was taken for the stent extra orally. These two scans were then superimposed to create an implant plan and construct stereolithographic surgical guides. With the assistance of these stereolithographic surgical guides and submerged surgical technique, 4 dental implants (IS III Active Implant, Neo BioTech) were placed in the canines and premolars regions of the maxillary arch, and 2 dental implants were placed in the canines region of the mandibular arch.

Each participants instructed to take Prophylactic broad spectrum antibiotic (875mg Amoxicillin and Clavulanic acid 125 mg) one hour before the surgery and for 7 days and rinsed their mouth with an antiseptic mouthwash (2% chlorohexidine) for 2 weeks after surgery. Additionally, non-steroidal anti-inflammatory drug (Diclofenac tablet 50 mg) was prescribed to control postoperative pain. One week after the surgery, the dentures were relived and relined with soft liner material (Mucosoft, Parkell, Edgewood. USA) and delivered to the participants. Follow-up visits were scheduled.

After the osseointegration period (3 months for the mandibular arch and 6 months for the maxillary arch), locator attachments (Neo Bio Tech) were screwed to the implants. Each patient received the following types of overdentures:

1. One mandibular implant-retained overdenture: After reliving the mandibular denture, direct pick-up technique was used to incorporate the attachments housing into the fitting surface of the mandibular denture.
2. Two designs of MaxIODs:

   * Conventional MaxIOD: After relieving the conventional maxillary denture, direct pick-up technique was used to incorporate the attachments housing into the fitting surface of the conventional maxillary denture.
   * Palateless MaxIOD: The conventional maxillary denture was duplicated and the palatal part was cut out, finished, and polished. The fitting surface was relived and direct pick-up technique was used to incorporate the attachments housing into the fitting surface of the palateless maxillary denture.

The participants were randomly allocated into two equal groups (7 per group). Randomization process was carried out by an independent examiner using a computer program, specifically Microsoft Excel. The first group of 7 participants received conventional MaxIODs. After a period of three months, the TOMASS test was done. Following this, they wore a palatless MaxIODs for an additional 3 months, after which the test was repeated. The second group of 7 patients initially received palatless MaxIODs. After three months of use, the TOMASS test was done. They then received conventional MaxIODs and the test was repeated after an additional three months. This randomization process was implemented in order to minimize the effect of the order of restoration on the measurements of swallowing threshold and efficiency.

Swallowing assessment:

TOMASS test was utilized to assess participants' swallowing abilities. (30) For this study, a commercially available cracker biscuit was used. Participants were instructed to sit on a chair in upright position and to eat the biscuit comfortably and as quickly as possible. They were also asked to say their name out loud as it indicate that they had finished the test. Using a video recorder the procedure was recorded for further analysis.

The recorded videos were then analyzed using the Avidemux 2.6 program to measure the following:

1. Swallowing threshold, which is the duration of chewing until the first swallow (determined by the moment of laryngeal elevation)
2. The TOMASS test parameters:

   1. Number of bites: The number of discrete bites taken to finish the cracker
   2. Number of masticatory cycles: As each cyclical mandibular movement up-down
   3. Number of swallows: As each vertical movement of the thyroid cartilage
   4. Total ingestion time: The time taken to complete the ingestion of the cracker from the first bite to the last.

ELIGIBILITY:
Inclusion Criteria:

* patient had sufficient bone quantity in the area between the mental foramina, sufficient inter-arch space, normal maxilla-mandibular relation, and have been edentulous for at least one year

Exclusion Criteria:

* Patients with uncontrolled systemic diseases, parafunctional habits, temporomandibular joint disorders, and a history of head/neck surgery were excluded, as were smoking and those who undergo radiation therapy.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
swallowing evaluation | after 3 months of overdenture insertion
  TOMASS test was utilized to assess participants' swallowing abilities

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Mohammed Ibrahim, PhD, Principal Investigator — Mansoura university, Faculty of dentistry, prosthodontics department
Locations (1):
- faculty of dentistry, mansoura university Mansoura, Egypt,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karlsson F, Lovric L, Matthelie J, Brage L, Hagglund P. A Within-Subject Comparison of Face-to-Face and Telemedicine Screening Using the Timed Water Swallow Test (TWST) and the Test of Mastication and Swallowing of Solids (TOMASS). Dysphagia. 2023 Feb;38(1):483-490. doi: 10.1007/s00455-022-10490-w. Epub 2022 Jul 9. PMID 35809097